CLINICAL TRIAL: NCT01770145
Title: A Phase 4, Open-Label, Efficacy and Safety Study of Apokyn® for Rapid and Reliable Improvement of Motor Symptoms in Parkinson Disease Subjects With Delayed Onset of L-Dopa Action
Brief Title: Apokyn for Motor IMProvement of Morning AKinesia Trial (AM IMPAKT)
Acronym: AM IMPAKT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MDD US Operations, LLC a subsidiary of Supernus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Supernus Pharmaceuticals, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USWM-AP1-4001
Record Dates: First submitted 2013-01-07; First posted 2013-01-17 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2017-10

CONDITIONS: Parkinson's Disease; Motor Symptoms; Akinesia; Hypomobility; Delayed Levodopa Onset
Keywords: Motor symptoms; Parkinson's Disease; Delayed Onset; Akinesia; Hypomobility; Unified Parkinson Disease Rating Scale (UPDRS) motor scores; Dopamine agonist; Apomorphine; Apokyn; Levodopa
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine; Levodopa; Carbidopa; carbidopa, levodopa drug combination; trimethobenzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- APOKYN (Experimental): APOKYN (apomorphine hydrochloride injection) is used as needed to treat off-episode motor symptoms, such as muscle stiffness, slow movements, and difficulty starting movements, in people with advanced Parkinson's disease (PD).
  In the study, subjects will complete an L-Dopa Baseline Period in which they record daily "time to on" following their regularly scheduled L-Dopa morning dose for 7 days. At the end of the baseline period, patients will start trimethobenzamide therapy during a minimum 3-Day Anti-Emetic Pretreatment Period. Patients determined to remain eligible at the end of the required Anti-Emetic Pretreatment Period will be initiated on APOKYN therapy by an investigator. Once the appropriate dose is identified by a study investigator, patients will inject APOKYN at their regularly scheduled levodopa morning dose time (levodopa will be delayed by 40 minutes) daily during a 7-day APOKYN Treatment Period and record "time to on" following the APOKYN injection.
  Interventions: Drug: APOKYN; Drug: L-dopa; Drug: Trimethobenzamide

INTERVENTIONS:
Drug: APOKYN — Apokyn will be titrated to an optimum dose which reproduces 90% of the subjects' "best on" UPDRS score during the Initiation Period. During the APOKYN Treatment Period, subjects will inject the dose identified in the initiation period once daily at the time of their normal scheduled L-Dopa dose (L-Dopa will be delayed by 40 minutes).
  Other Names: apomorphine hydrochloride injection
Drug: L-dopa — Subjects on a stable L-Dopa regimen will be entered into the study. For the L-Dopa Baseline Period through the Initiation Period, subjects will continue their normal L-Dopa dosing regimen. During the APOKYN Treatment Period, subjects will replace their normally scheduled first morning L-Dopa dose with an APOKYN injection, and then administer their normal first morning L-Dopa dose 40 minutes later.
  Other Names: Levodopa, Levodopa/Carbidopa, Sinemet, Sinemet CR, Parcopa
Drug: Trimethobenzamide — Following the L-Dopa Baseline Period, subjects will initiate trimethobenzamide treatment TID for a minimum of 3 days during a Anti-Emetic Pretreatment Period. Subjects will continue trimethobenzamide therapy TID through the duration of the APOKYN Initiation Period and APOKYN Treatment Period.
  Other Names: Tigan

SUMMARY:
This study is designed to assess the effect of APOKYN treatment in rapid and reliable improvement of motor symptoms in Parkinson's disease (PD) subjects suffering from delayed or unreliable onset of levodopa (L-dopa) action.

DETAILED DESCRIPTION:
This Phase IV, Open-Label, Efficacy and Safety Study of APOKYN® is intended to assess the effect of APOKYN treatment in rapid and reliable improvement of motor symptoms in PD subjects suffering from delayed or unreliable onset of L-dopa action. The study will also include a sub-group of 8 subjects to evaluate their gastroparesis and assess their gastric empty with other measures to explore if APOKYN has any influence on gastric empty rather than just bypassing the stomach with a subcutaneous route of administration.

The primary objective of this study is to assess the effect of APOKYN treatment in rapid and reliable improvement of motor symptoms in PD subjects suffering from delayed or unreliable onset of L-dopa action (defined below). APOKYN treatment will also be assessed in a sub-group of PD subjects suffering from gastroparesis and delayed onset of L-dopa action.

Delayed or unreliable onset to L-dopa for the study population is defined as impaired motor function (tremor, bradykinesia, rigidity, and/or postural instability) persisting for a minimum of 45 minutes after taking a dose of L-dopa because of its delay in onset of action. The impaired motor function resulting from delay in L-dopa onset is referred to as "delayed ON" and when it occurs upon awakening is referred to as "morning akinesia."

Main Study:

This is a multicenter, multiple-treatment, open-label, outpatient study to evaluate the efficacy and safety of APOKYN in PD subjects with delayed onset of L dopa action. The study will have:

* Screening - 1-5 days (Visit 1);
* Baseline L-Dopa Period - 7 days, continuation of L dopa treatment;
* Antiemetic Treatment Period - 3-days; initiation of trimethobenzamide 300 mg tid orally;
* APOKYN Initiation/optimum dose identification Period (Visit 2)- variable, not more than 11 days;
* APOKYN Treatment Period - 7 days, immediately upon identification of optimum dose;
* Study Discharge (Visit 3)- within 2 days of completion of the APOKYN treatment period.

Gastroparesis Sub-Study:

A sub-group of subjects (n=8) from 1 study site that have symptoms of gastroparesis will be admitted to the clinic on 2 occasions to undergo gastroparesis procedures and assessments (once at the conclusion of the baseline L-dopa period and once at the conclusion of the APOKYN treatment period). Note, to do the second gastroparesis assessment, this sub-group of subjects will have an extension for one extra day beyond the designated 7 day APOKYN treatment period (i.e., it will be 8 days) in order to keep the 7 day diary recording outpatient scope of work the same as the rest of the subjects in the study. The second inpatient period will be also considered the end-of-study visit for this sub group.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age.
2. Idiopathic PD.
3. Not currently taking APOKYN and, if previously prescribed APOKYN, did not discontinue therapy due to intolerable side effects/safety reasons.
4. Prescribed L-dopa therapy at a steady maintenance dose, representing an optimal treatment regimen in the opinion of the Investigator, for at least 4 weeks before study participation.
5. Minimum subject-reported time to turn "on" (TTO) in the early morning (time to end akinetic/ bradykinetic state resulting from delay in L-dopa onset of action) of 45 minutes after the first morning L-dopa dose for a minimum of 3 days/week (as determined with the subject diary at Visit 2).
6. Able to adequately differentiate between and describe variations in "on" and "off" states in the opinion of the Investigator.
7. I to III Modified Hoehn and Yahr stage in the "on" state (Appendix B).
8. Be seeking treatment for early morning akinesia.
9. If female and of childbearing potential, must agree to use one of the following methods of birth control:

   * Oral contraceptive;
   * Patch;
   * Barrier (diaphragm, sponge or condom) plus spermicidal preparations;
   * Intrauterine contraceptive system;
   * Levonorgestrel implant;
   * Medroxyprogesterone acetate contraceptive injection;
   * Complete abstinence from sexual intercourse;
   * Hormonal vaginal contraceptive ring; or
   * Surgical sterilization or partner sterile (must have documented proof).
10. Access to a live-in caregiver, if needed.
11. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study-related procedures to complete the study.
12. Able to verbalize understanding of the consent form, able to provide written informed consent.

    The following must be present for inclusion in the single site gastroparesis sub-study:
13. Have symptoms of gastroparesis.
14. Have improvement of at least one Modified Hoehn and Yahr stage from "off" to "on."
15. Currently seeking treatment for delayed L-dopa onset.
16. Have no allergy to eggs.

Exclusion Criteria:

1. Changes in L-dopa dosing regimen 4 weeks before the screening visit.
2. Female who is pregnant or lactating.
3. Contraindications to APOKYN or hypersensitive to apomorphine hydrochloride or any of the ingredients of APOKYN (notably sodium metabisulfite).
4. Participation in any other clinical trial within 14 days of the screening visit.
5. Receipt of any investigational (i.e., unapproved) medication within 30 days of the screening visit.
6. Currently taking, or likely to need to take at any time during the course of the study, any 5HT3 antagonist (i.e., ondansetron, granisetron, dolasetron, palonosetron, alosetron).
7. Currently taking medications for treatment of gastroparesis (e.g., erythromycin, cisapride, metoclopramide).
8. Malignant melanoma or a history of previously treated malignant melanoma within 5 years.
9. Serious medical illness including, but not limited to:

   * Liver disease;
   * Kidney problems; and
   * Heart problems.
10. Psychiatric disorder, including but not limited to dementia or any disorder that, in the opinion of the Investigator requires ongoing treatment that would make study participation unsafe or make treatment compliance difficult.
11. Lack of compliance and follow-up.
12. Any other condition, current therapy, or prior therapy (within 30 days of the screening visit), which, in the opinion of the Investigator, would make the subject unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2012-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianpiera H. Ceresoli-Borroni, PhD, Study Director — Supernus Pharmaceuticals
Locations (12):
- United States (12):
  - Keck School of Medicine, Los Angeles, California
  - Neurosearch, Inc., Reseda, California
  - Georgetown University, Washington D.C., District of Columbia
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Henry Ford West Bloomfield Hospital, Bloomfield Hills, Michigan
  - Parkinson's Disease and Movement Disorders Center of New York, Commack, New York
  - University of Cincinnati Academic Health Center, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - University of Texas Health Science Center, Houston, Department of Neurology, Houston, Texas
  - Center for Neurological Care and Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- APOKYN: Subjects will complete an L-Dopa Baseline Period in which they record daily "time to on" following their regularly scheduled L-Dopa morning dose for 7 days. At the end of the baseline period, patients will start trimethobenzamide therapy during a minimum 3-Day Anti-Emetic Pretreatment Period. Patients determined to remain eligible at the end of the required Anti-Emetic Pretreatment Period will be initiated on APOKYN therapy by an investigator. Once the appropriate dose is identified by a study investigator, patients will inject APOKYN at their regularly scheduled levodopa morning dose time (levodopa will be delayed by 40 minutes) daily during a 7-day APOKYN Treatment Period and record "time to on" following the APOKYN injection.
Period: Baseline
Arm/Group | APOKYN
Started | 127
Completed | 101
Not Completed | 26
Not completed — Adverse Event | 20
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1
Not completed — Unable to define optimal dose | 4
Period: Treatment
Arm/Group | APOKYN
Started | 101
Completed | 97
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | APOKYN
Number analyzed (Participants) | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.20 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 84
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 121
  Hispanic or Latino | 6
Duration of Parkinson's Disease (years) [Number; unit: participants]
  0-5 years | 21
  6-10 years | 48
  11-15 years | 34
  15+ years | 24
Duration of Akinesia (years) [Number; unit: participants]
  <2 years | 44
  2-4 years | 35
  5-6 years | 16
  >6 years | 28
  Unknown | 4
Average Daily Time to On [Mean (Standard Deviation); unit: minutes] | 59.13 (18.13)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily "Time to on" ("TTO") by Subject Diary.
Description: Patients will record daily "time to on" or "TTO" following their regularly scheduled first L-Dopa dose in the baseline period for 7 consecutive days. Following initiation on Apokyn therapy, patients will inject Apokyn at their regularly scheduled L-Dopa time (L-Dopa dosing will be delayed by 40 minutes following Apokyn injection) and record "time to on" or "TTO" from the injection. "Time to on" for both periods will be recorded in a standardized subject diary. Daily "TTO" for the baseline period will be averaged for each subject and compared to the daily "TTO" for the same subject during the treatment period to assess APOKYN's effect on "TTO".
Time Frame: L-Dopa Baseline Days 1-7 and APOKYN Treatment Days 1-7
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- APOKYN: In the study, subjects will complete an L-Dopa Baseline Period in which they record daily "time to on" following their regularly scheduled L-Dopa morning dose for 7 days. At the end of the baseline period, patients will start trimethobenzamide therapy during a minimum 3-Day Anti-Emetic Pretreatment Period. Patients determined to remain eligible at the end of the required Anti-Emetic Pretreatment Period will be initiated on APOKYN therapy by an investigator. Once the appropriate dose is identified by a study investigator, patients will inject APOKYN at their regularly scheduled levodopa morning dose time (levodopa will be delayed by 40 minutes) daily during a 7-day APOKYN Treatment Period and record "time to on" following the APOKYN injection.
Arm/Group | APOKYN
Number analyzed (Participants) | 88
minutes
  Baseline | 60.86 (18.11)
  Treatment Period | 23.72 (14.55)
  Change from Baseline | 37.14 (20.51)

2. Secondary Outcome: Change From Baseline in Gastric Emptying Time
Description: A sub-group of subjects from 1 study site that have symptoms of gastroparesis were admitted to the clinic on 2 occasions to undergo gastroparesis procedures and assessments (once at the conclusion of the baseline L-dopa period and once at the conclusion of the APOKYN treatment period). Note, to do the second gastroparesis assessment, this sub-group of subjects had an extension for one extra day beyond the designated 7 day APOKYN treatment period (i.e., it will be 8 days) in order to keep the 7 day diary recording outpatient scope of work the same as the rest of the subjects in the study. The second inpatient period was also considered the end-of-study visit for this sub group.
Time Frame: L-Dopa Baseline Days 1-7 and APOKYN Treatment Days 1-8
Population: A sub-group of subjects from 1 study site that have symptoms of gastroparesis were admitted to the clinic to undergo gastroparesis procedures and assessments (once at the conclusion of the baseline L-dopa period and once at the conclusion of the APOKYN treatment period)
Arm/Group | APOKYN
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | APOKYN
Serious Adverse Events (participants affected / at risk) | 0/127
Other Adverse Events (participants affected / at risk) | 70/127
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APOKYN (N=127)
Chills (General disorders) | 6 (6)
Chest Pain (General disorders) | 1 (1)
Chest Discomfort (General disorders) | 2 (2)
Vomiting (General disorders) | 6 (6)
Toothache (Gastrointestinal disorders) | 1 (1)
Salivary hyper-secretion (Gastrointestinal disorders) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 25 (25)
Diarrhea (Gastrointestinal disorders) | 0 (0)
Vision blurred (Eye disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Eyelid ptosis (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Tooth Injury (Injury, poisoning and procedural complications) | 0 (0)
Stress Fracture (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0)
Joint Sprain (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Tooth Infection (Infections and infestations) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0)
Oedema (General disorders) | 2 (2)
Injection Site Pruritus (General disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (1)
Injection site bruising (General disorders) | 0 (0)
Feeling hot (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0)
Syncope (Nervous system disorders) | 0 (0)
Somnolence (Nervous system disorders) | 7 (7)
Paraesthesia (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0)
Hyposaethesia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Dyskinesia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Heart rate increased (Investigations) | 1 (1)
Pallor (Vascular disorders) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 0 (0)
Hot flush (Vascular disorders) | 1 (1)
Flushing (Vascular disorders) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1)
Yawning (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Sneezing (Skin and subcutaneous tissue disorders) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Full analysis set (n=88) included patients who completed 5/7 days of diary entries in APOKYN treatment period. The gastroparesis sub-study to assess prevalence and severity of gastroparesis was not analyzed because too few subjects were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor shall have the first right, within nine months following the Sponsor having in its possession all data related to the Study, to publish the Study lead paper. Following the foregoing, the Institution shall have the right, consistent with academic standards, to publish the results of Study provided the Institution provides a publications committee, comprised of at least the Sponsor, with a draft at least thirty (30) days prior to planned submission.